CLINICAL TRIAL: NCT03290898
Title: REPLACE: Can Exercise Replace Inhaled Corticosteroid Treatment in Asthma? A Randomized Clinical Trial
Brief Title: REPLACE: Can Exercise Replace Inhaled Corticosteroid Treatment in Asthma? A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Backer, Professor dr.med., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REPLACE
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: Asthma; Exercise; Asthma treatment; Inhaled corticosteroid; Rehabilitation
MeSH Terms: conditions — Asthma; Motor Activity | interventions — High-Intensity Interval Training; Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: A randomized, controlled parallel group, outcome assessor blinded, clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blindet, randomization and training intervention by non-investigator. Open-label after primary follow up. After unblinding, blindet 3rd party performs tests (visit 9 and 12 months, e.g. spirometry)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): Supervised High intensity interval training (HIIT) 3 times a week for 6 months.
  Training session:
  10 minutes warm up (Low-moderate intensity) 30 minutes intervention (16 minutes HIIT) 10 minutes cool down(Low-moderate intensity)
  Interventions: Behavioral: High Intensity Interval Training
- Control group (No Intervention): Control group, usual lifestyle. Aside from training intervention, all other visits are the same as intervention group (training).

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Training (HIIT)
  Other Names: Training group
  Arms: Training group

SUMMARY:
To evaluate if physical exercise intervention leads to an improved asthma control as measured by Asthma Control Questionnaire (ACQ-5) in such a magnitude that inhaled corticosteroid can be reduces in asthmatics.

DETAILED DESCRIPTION:
At least 102 asthmatics will be randomized 2:1 (2 to training group; 1 to control) and undergo 6 months of intervention or usual lifestyle.

Subjects must have confirmed asthma diagnosis, on a stable treatment with inhaled corticosteroid, symptomatic and untrained.

At enrollment and during the study asthma medicine is adjusted based on asthma symptoms evaluated by ACQ-5. 6 treatment steps are pre-defined, and if well controlled asthma, subjects are down-titrated one step, if uncontrolled, subjects are uptitrated one step.

ELIGIBILITY:
Inclusion Criteria:

* Asthma (The diagnose of asthma is based on symptoms and at least one positive asthma test the last 5 years (AHR to either mannitol or methacholine, reversibility to beta2-agonist, peak flow variation or positive eucapnic voluntary hyperventilation test))
* ACQ ≥ 1 and ≤ 2.5
* On a daily dose of ICS at a minimum of 400 µg budesonide or equivalent ICS for 3 months and with no changes in asthma medicine 4 weeks prior to enrollment
* Untrained (no participation in vigorous exercise for more than 1 hour per week during the last 2 month)
* Capable of exercising on bike

Exclusion Criteria:

* Unable to speak and understand Danish
* Infection within 4 weeks prior to visit 100*
* Asthma exacerbation within 4 weeks prior to visit 100*
* Hospitalized for an asthma attack during the last 2 months
* Treatment with immunotherapy within 5 T½ of the treatment drug prior to visit 100
* Initiation of allergen immunotherapy within 3 months prior to visit 100 or plan to begin therapy during study period
* Treatment with peroral prednisolone
* Respiratory: other chronic pulmonary disease of clinically significance
* Cardiovascular: Unstable ischemic heart disease, myocardial infarction within the last 12 months, symptomatic heart failure (NYHA III-IV or EF <40%), symptomatic heart arrhythmia (documented with ECG), uncontrolled hypertension (>155/100)
* Pregnancy or breastfeeding or planned pregnancy within the next 12 months
* Other inflammatory or metabolic diseases with the exception of rhinitis, atopy and well-controlled hypothyroidism treated with or without Eltroxin
* Vaccination less than 2 weeks prior to any visit
* Current or former smokers with > 20 pack years
* Subjects, who by investigators determination, will not be able to adhere to study protocol

  * If patients are excluded due to a recent infection or exacerbation they can undergo re-screening after a total of 4 weeks after end of exacerbation treatment/clearing the infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Reduced inhaled corticosteroid (ICS) 6 months | 6 months +/- 7 days
  The proportion of participants at 6 months that have been down-titrated in ICS dose by at least 25% compared to the participants' baseline dose

SECONDARY OUTCOMES:
Reduced inhaled corticosteroid (ICS) 12 months | 12 months +/- 7 days
  The proportion of participants at 12 months that have been down-titrated in ICS dose by at least 25 % compared to baseline.
Cumulated ICS 6 months | 6 months +/- 7 days
  Change from baseline in cumulated dose of ICS at 6 months
Cumulated ICS 12 months | 12 months +/- 7 days
  Change from baseline in cumulated dose of ICS at 12 months
Cumulated Long acting beta2 agonists (LABA) 6 months | 6 months +/- 7 days
  Change from baseline in cumulated dose of LABA at 6 months
Cumulated LABA 12 months | 12 months +/- 7 days
  Change from baseline in cumulated dose of LABA at 12 months
Exacerbation rate 6 months | 6 months +/- 7 days
  Number of exacerbations (moderate-severe) at 6 months
Exacerbation rate 12 months | 12 months +/- 7 days
  Number of exacerbations (moderate-severe) at 12 months
miniAQLQ 6 months | 6 months +/- 7 days
  Change from baseline in Asthma life quality evaluated by miniAQLQ at 6 months
miniAQLQ 12 months | 12 months +/- 7 days
  Change from baseline in Asthma life quality evaluated by miniAQLQ at 12 months
Fraction of exhaled Nitrogen Oxid 6 months | 6 months +/- 7 days
  Change from baseline in Airway inflammation evaluated by FeNO at 6 months
Fraction of exhaled Nitrogen Oxid 12 months | 12 months +/- 7 days
  Change from baseline in Airway inflammation evaluated by FeNO at 12 months
Sputum cell count 6 months | 6 months +/- 7 days
  Change from baseline in Airway inflammation evaluated by sputum cell count at 6 months
Sputum cell count 12 months | 12 months +/- 7 days
  Change from baseline in Airway inflammation evaluated by sputum cell count at 12 months
Systemic inflammation 6 months | 6 months +/- 7 days
  Change from baseline in systemic inflammation evaluated by blood eosinophilic, hsCRP and inflammatory cytokines (e.g. IL-6 and IL-8) and TNF-alfa at 6 months
Systemic inflammation 12 months | 12 months +/- 7 days
  Change from baseline in systemic inflammation evaluated by blood eosinophilic, hsCRP and inflammatory cytokines (e.g. IL-6 and IL-8) and TNF-alfa at 12 months
Airway hyperresponsiveness | 6 months +/- 7 days
  Change from baseline in airway hyperresponsiveness measured by methacholine test at 6 months
FEV1 6 months | 6 months +/- 7 days
  Change from baseline in lung function evaluated by FEV1 at 6 months
FVC 6 months | 6 months +/- 7 days
  Change from baseline in lung function evaluated by FVC at 6 months
FEV1 12 months | 12 months +/- 7 days
  Change from baseline in lung function evaluated by FEV1 at 12 months
FVC 12 months | 12 months +/- 7 days
  Change from baseline in lung function evaluated by FVC at 12 months
Cardiopulmonary fitness | 6 months +/- 7 days
  Change from baseline in cardiopulmonary fitness evaluated by maximum oxygen consumption at 6 months (VO2max)
Change in fat and muscle composition (DEXA scan) | 6 months +/- 7 days
  Change from baseline in fat and muscle composition evaluated by DEXA scan

OTHER OUTCOMES:
Eosinophilic subpopulation - exploratory analyses 6 months | 6 months +/- 7 days
  To evaluate the effect of the intervention in sub-populations of asthmatics using different cut-off values of blood eosinophilics. Both regarding primary outcome and secondary outcomes.
Eosinophilic subpopulation - exploratory analyses 12 months | 12 months +/- 7 days
  To evaluate the effect of the intervention in sub-populations of asthmatics using different cut-off values of blood eosinophilics with regards to secondary outcomes at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Respiratory Research Unit, Birpebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitzner-Fabricius A, Dall CH, Henriksen M, Hansen ESH, Toennesen LL, Hostrup M, Backer V. Effect of High-Intensity Interval Training on Inhaled Corticosteroid Dose in Asthma Patients: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2023 Jul;11(7):2133-2143.e8. doi: 10.1016/j.jaip.2023.04.013. Epub 2023 May 31. PMID 37256238

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03290898/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03290898/SAP_001.pdf